CLINICAL TRIAL: NCT00862394
Title: A 12-week, Multinational, Randomised, Double Blind, Double Dummy, 4-arm Parallel-group Study Comparing the Efficacy and Safety of CHF 1535 (Fixed Combination of Beclomethasone Dipropionate + Formoterol Fumarate) 100 + 6 μg/Actuation Inhalation Powder, Administered Via the NEXT Inhaler, Versus CHF 1535 (Fixed Combination of Beclomethasone Dipropionate + Formoterol Fumarate) 100 + 6 μg/Actuation, Via HFA Pressurised Inhalation Solution, in Moderate to Severe Symptomatic Asthmatic Patients Aged ≥ 12 Years Under Treatment With Inhaled Corticosteroids
Brief Title: A Study Comparing the Efficacy and Safety of CHF 1535 (BDP +FF) Inhalation Powder, Administered Via the NEXT Inhaler, Versus CHF 1535 (BDP +FF), Administered Via a pMDI, in Moderate to Severe Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CCD-0705-PR-0027
Record Dates: First submitted 2009-03-13; First posted 2009-03-16 (Estimated); Last update posted 2018-04-13 (Actual); Status verified 2018-04

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Foster Home Care

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): CHF 1535 Next DPI : BDP/Formoterol : 200/12 µg
  Interventions: Drug: BDP/Formoterol Next DPI
- 2 (Active Comparator): CHF 1535 HFA pMDI : BDP/Formoterol : 200/12 µg
  Interventions: Drug: Foster
- 3 (Experimental): CHF 1535 Next DPI : BDP/Formoterol : 400/24 µg
  Interventions: Drug: BDP/Formoterol Next DPI
- 4 (Active Comparator): CHF 1535 HFA pMDI : BDP/Formoterol : 400/24 µg
  Interventions: Drug: Foster

INTERVENTIONS:
Drug: BDP/Formoterol Next DPI — BDP/Formoterol Next DPI 100/6 µg (daily dose : 200/12 µg)
  Arms: 1
Drug: Foster — BDP/Formoterol HFA pMDI 100/6 µg (daily dose : 200/12 µg)
  Arms: 2
Drug: BDP/Formoterol Next DPI — BDP/Formoterol 100/6 µg (daily dose : 400/24 µg)
  Arms: 3
Drug: Foster — BDP/Formoterol HFA pMDI 100/6 µg (daily dose : 400/24 µg)
  Arms: 4

SUMMARY:
To demonstrate that CHF 1535 via NEXT DPI (beclomethasone dipropionate + formoterol fumarate 100 + 6 μg), 1 inhalation or 2 inhalations twice daily, for 12 weeks is non-inferior to the corresponding dose of CHF 1535 via HFA-134a "extrafine" pMDI in terms of pulmonary function in moderate to severe symptomatic asthmatic patients aged ≥ 12 years under treatment with inhaled corticosteroids

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Outpatients of both sexes, aged > 12 years
* Moderate to severe symptomatic asthma
* Forced expiratory volume in the first second (FEV1) > 40% and < 80% of the predicted normal values
* Reversibility test
* "Partly controlled" asthma (GINA revised 2006)
* Patients free of long-acting beta2-agonists (LABAs) treatment
* Under inhaled corticosteroids (ICS) treatment
* A minimum inspiratory flow ≥ 40 L/min 10.
* Non-smokers or ex smokers
* Asthma Control Questionnaire ACQ score ≥ 1.5

Exclusion Criteria:

* Pregnant or nursing (lactating) women
* Women of child-bearing potential, UNLESS they are menopausal or have acceptable methods of contraception
* Significant seasonal variation in asthma or asthma occurring only during episodic exposure to an allergen or a chemical sensitizer
* History of near fatal asthma
* Occurrence of asthma exacerbations or respiratory tract infections in the 6 weeks preceding the screening visit
* Diagnosis COPD
* History of cystic fibrosis, bronchiectasis or alpha-1 antitrypsin deficiency
* Diagnosis of restrictive lung disease
* Patients treated with oral or parenteral corticosteroids in the previous 2 months (3 months for parenteral depot corticosteroids)
* Intolerance or contra-indication to treatment with beta2-agonists and/or inhaled corticosteroids
* Allergy to any component of the study treatments
* Any change in the dose, schedule, formulation or product of an inhaled corticosteroid in the 4 weeks prior to screening visit
* Significant medical history of and/or treatments for cardiac, renal, neurological, hepatic, endocrine diseases, or any laboratory abnormality ;
* Patients with abnormal QTc

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 783 (Actual)
Dates: Start 2009-02; Primary Completion 2009-10 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline measured at clinic to the end of treatment period in pre-dose morning FEV1 (L) measured at clinic | 3 month period

SECONDARY OUTCOMES:
Pre-dose FEV1 | every month
Post-dose FEV1 AUC 0-8 h | 3 month period
FVC and FEF 25-75% | every month
PEF | every day
Morning and evening asthma clinical symptoms scores | every day
Moderate and severe exacerbations | every month
Rescue medication | every day
Sputum | 3 month period

CONTACTS AND LOCATIONS:
Locations (1):
- Oliver Kornmann - National Coordinator in Germany, Mainz, Germany

REFERENCES:
- See also: Study Record on EU Clinical Trials Register including results — https://www.clinicaltrialsregister.eu/ctr-search/search?query=CCD-0705-PR-0027